CLINICAL TRIAL: NCT02820259
Title: Therapeutic Drug Monitoring of Tacrolimus Biliary Concentrations for Liver-transplanted Patients (STABILE)
Acronym: STABILE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_9755
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Biliary Concentration of Tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
The purpose of this study is to demonstrate that the biliary concentration of TCR is a good marker of its immunosuppressive activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years) of both sexes,
* Candidates for liver transplantation or retransplantation, whatever the etiology and severity of the underlying disease,
* Not having expressed their opposition to participation in the study

Exclusion Criteria:

* Bilio-enteric anastomosis,
* Associated transplantation of another organ
* Contraindications to TCR administration
* Delayed introduction of TCR (beyond the 5th postoperative day) whatever the cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver-transplanted patients who receive tacrolimus
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-05-01; Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
coefficient of correlation (r²) between the biliary concentration of TCR and concentration within PBMC | during the first 7 days after its initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Rennes, Rennes, France

REFERENCES:
- [Derived] Rayar M, Tron C, Locher C, Chebaro A, Beaurepaire JM, Blondeau M, Cusumano C, Bardou-Jacquet E, Houssel-Debry P, Camus C, Petitcollin A, Verdier MC, Lakehal M, Desfourneaux V, Sulpice L, Meunier B, Bellissant E, Boudjema K, Lemaitre F. Tacrolimus Concentrations Measured in Excreted Bile in Liver Transplant Recipients: The STABILE Study. Clin Ther. 2018 Dec;40(12):2088-2098. doi: 10.1016/j.clinthera.2018.10.015. Epub 2018 Nov 19. PMID 30467013